CLINICAL TRIAL: NCT04702191
Title: Promoting Healthy Families: A Canadian Evaluation of Two Evidence-based Parenting Programs
Brief Title: Promoting Healthy Families: A Canadian Evaluation
Acronym: PHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of Manitoba (Other); Institute for Clinical Evaluative Sciences (Other); Public Health Agency of Canada (PHAC) (Other Government); University of Exeter (Other)
Responsible Party: Principal Investigator, Andrea Gonzalez (for Nathan), Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10583
Record Dates: First submitted 2021-01-02; First posted 2021-01-08 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Child Behavior Problem; Parenting
Keywords: child behavior problem, parenting, parental capacity
MeSH Terms: interventions — (tris(diphenylphosphinomethyl)phenylborate)(p-tolylnitrido)iron(I)

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triple P (Positive Parenting Program) (Experimental): Triple P - level 4 group: All 600 participants will undergo screening and a baseline assessment before randomization. Once randomized, the Triple P group (n=200) will be provided with 8-week group/individual sessions.
  Interventions: Behavioral: Triple P
- Circle of Security Parenting (Experimental): Circle of Security - Parenting (COS-P): Once randomized to the COSP group (n=200), caregivers will be provided with an 8-week group session.
  Interventions: Behavioral: Circle of Security Parenting
- Treatment As Usual (No Intervention): Treatment as usual: Caregivers randomized to this arm (n=200) will receive either a different program, or brief services depending on the organization.

INTERVENTIONS:
Behavioral: Triple P — Triple P - level 4 group is a group-based parenting intervention for families with children who exhibit behavioural or emotional difficulties. Group sessions typically focus on topics such as positive parenting, helping children develop, managing misbehaviour, and planning ahead. Practitioners then provide individual feedback on progress using positive parenting strategies and goal setting. Trained practitioners will deliver the program according to the manualized protocol (Turner, Markie-Dadds, & Sanders, 2010). This will include eight weekly sessions with maximum of 12 parents. The first four sessions will be as group sessions. These four group sessions will be followed by three one-to-one practical and personalised telephone consultations. Finally, there will be one group session, which will complete the programme and parents' contact with the Triple P practitioners. The main aim of this session is to review progress and plan for the future.
  Other Names: Triple P - group level 4
  Arms: Triple P (Positive Parenting Program)
Behavioral: Circle of Security Parenting — Circle of Security - Parenting (COS-P) will be delivered according to the protocol outlined by Cooper, Hoffman and Powell (Cooper et al., 2009). COS-P is a manualized eight-session parent-education group program which has the same broad aims and core components of the COS-Intensive model from which it was developed (i.e., to increase caregiver sensitivity and responsiveness to child cues, empathy for the child by supporting parental reflective functioning, recognition and understanding of child attachment cues, and awareness of the impact of the caregiver's own attachment history on caregiving patterns). The program is led by one or two facilitators and includes 10-12 caregivers. The program uses clinical DVD clips of problematic parent-child interaction and healthy alternatives to illustrate attachment patterns and parenting styles, and to promote group discussion.
  Arms: Circle of Security Parenting

SUMMARY:
Interventions that promote safe, stable, and nurturing relationships between caregivers and children are key to improving healthy family relationships, reducing child socioemotional and behaviour problems, and preventing child maltreatment. Although a broad range of parenting programs are currently implemented in communities across Ontario, most programs are inadequately evaluated, or else not evaluated at all. Using a three-armed randomized controlled trial, the aim of the current study is to evaluate the effectiveness of two parenting programs, the Triple P - Positive Parenting Program (group - level 4) and the Circle of Security Parenting Program (group) compared to treatment as usual in Ontario, Canada.

DETAILED DESCRIPTION:
The overall goal of the evaluation is to provide robust evidence about the implementation and effectiveness of two parenting programs, the Triple P and Circle of Security Parenting (COSP), in the province of Ontario, on parenting practices and functioning, and child emotional behaviour problems outcomes, and secondary outcomes including selected child maltreatment-related outcomes. These objectives will be achieved in two phases. The investigators will conduct a multi-site, three-arm randomized controlled trial of 600 participating caregivers and their children to compare Triple P (level 4 group) and COSP to treatment as usual (TAU) with respect to improving positive practices and child outcomes. Participants will be randomly assigned to one of the three conditions using stratified (by site) block randomization. All participants will undergo screening and a baseline assessment before randomization. Once randomized, the Triple P and COSP caregivers will receive 8-week session. The TAU group will receive a different program, or short therapy sessions depending on the organization. Caregivers will complete follow-up assessments at post-treatment, 6- and 12-months.

ELIGIBILITY:
Inclusion Criteria:

Caregivers of children are eligible for inclusion if:

* Custodial caregiver of child is aged 2 to 6 years at time of screening.
* Families with sufficient knowledge of English needed for assessment measures.
* Caregivers capable of giving informed, written consent.
* Definition of 'at-risk' as measured by one of the following criteria as outlined below:

  * Elevated child emotional behavioural problems as indexed by above- population mean total scores on the Strengths and Difficulties Questionnaire (SDQ); OR
  * One of the following family or contextual risk factor
  * Parental challenge - parental mental health problems, as indexed by score on K6 distress scale ≥ 13; adolescent parent status (less than 20 years of age); single parent status; OR Sociodemographic risk factor - parent with less than grade 12 education; parent on social assistance;
  * Expressed difficulties with parenting: Do you often feel like your child is difficult to take care of?

Exclusion Criteria:

• Children with suspected severe to profound developmental delay.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 502 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-17 (Actual)

PRIMARY OUTCOMES:
Child emotional/behavioural problems | 6-months
  The investigators will measure change in child emotional and behavioural problems across time points.
Parenting Practices | 6-months
  Discipline style measured using the Parenting Scale

SECONDARY OUTCOMES:
Change in Observed Parenting | Baseline, 6-months.
  Video-taped caregiver-child interactions

OTHER OUTCOMES:
Caregiver Emotion Regulation | Baseline, 6- and 12-months.
  Change in Parental Emotional Regulation will be measured using the Difficulties in Emotion Regulation Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Gonzalez, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold, D.S., O'Leary, S.G., Wolff, L.S., & Acker, M.M. (1993). The Parenting Scale: A Measure of Dysfunctional Parenting in Discipline Situations. Psychological Assessment, 5(2), 137-144.
- [Background] Cooper, G., Hoffman, K., Powell, B., & Marvin, R. (2005). The circle of security intervention: Differential diagnosis and differential treatment. In L. J. Berlin, Y. Ziv, L. Amaya-Jackson, & M. T. Greenberg (Eds.), Enhancing early attachments: Theory, research, intervention, and policy (pp. 127-151). New York, NY: The Guilford Press.
- [Background] Cooper, G., Hoffman, K., & Powell, B. (2009). Circle of Security Parenting: A relationship based parenting program. Facilitator DVD Manual 5.0. Spokane, WA: Circle of Security International. Marycliff Institute.
- [Background] de Graaf I, Speetjens P, Smit F, de Wolff M, Tavecchio L. Effectiveness of the Triple P Positive Parenting Program on behavioral problems in children: a meta-analysis. Behav Modif. 2008 Sep;32(5):714-35. doi: 10.1177/0145445508317134. Epub 2008 May 12. PMID 18475003
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Hoffman KT, Marvin RS, Cooper G, Powell B. Changing toddlers' and preschoolers' attachment classifications: the Circle of Security intervention. J Consult Clin Psychol. 2006 Dec;74(6):1017-26. doi: 10.1037/0022-006X.74.6.1017. PMID 17154732
- [Background] Kaufman, E.A., Xia, M., Fosco, G. et al. (2016). The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and Replication in Adolescent and Adult Samples. Journal of Psychopathology and Behavioral Assessment, 38, 443-455 (2016).
- [Background] Marryat L, Thompson L, Wilson P. No evidence of whole population mental health impact of the Triple P parenting programme: findings from a routine dataset. BMC Pediatr. 2017 Jan 31;17(1):40. doi: 10.1186/s12887-017-0800-5. PMID 28143454
- [Background] Maxwell AM, McMahon C, Huber A, Hawkins E, Reay RE. Addressing the Evidence Gap: Protocol for an Effectiveness Study of Circle of Security Parenting, an Attachment-Based Intervention. Front Glob Womens Health. 2020 Oct 22;1:575752. doi: 10.3389/fgwh.2020.575752. eCollection 2020. PMID 34816157
- [Background] Public Health Agency of Canada (2016). Chief Public Health Officer of Canada. Report on the State of Public Health in Canada 2016: A Focus on Family Violence in Canada. Cat: HP2-1DE-PDF. ISSN: 1924-7087. Pub: 160152. Ottawa.
- [Background] Prinz RJ, Sanders MR, Shapiro CJ, Whitaker DJ, Lutzker JR. Population-based prevention of child maltreatment: the U.S. Triple p system population trial. Prev Sci. 2009 Mar;10(1):1-12. doi: 10.1007/s11121-009-0123-3. PMID 19160053
- [Background] Prinz RJ, Sanders MR, Shapiro CJ, Whitaker DJ, Lutzker JR. Erratum to: Population-Based Prevention of Child Maltreatment:The U.S. Triple P System Population Trial. Prev Sci. 2015 Jan;16(1):168. doi: 10.1007/s11121-014-0538-3. No abstract available. PMID 25483885
- [Background] Prinz RJ, Sanders MR, Shapiro CJ, Whitaker DJ, Lutzker JR. Addendum to "Population-Based Prevention of Child Maltreatment: The U.S. Triple P System Population Trial". Prev Sci. 2016 Apr;17(3):410-6. doi: 10.1007/s11121-016-0631-x. PMID 26780665
- [Background] Sanders MR, Ralph A, Sofronoff K, Gardiner P, Thompson R, Dwyer S, Bidwell K. Every family: a population approach to reducing behavioral and emotional problems in children making the transition to school. J Prim Prev. 2008 May;29(3):197-222. doi: 10.1007/s10935-008-0139-7. PMID 18461457
- [Background] Sanders MR. Development, evaluation, and multinational dissemination of the triple P-Positive Parenting Program. Annu Rev Clin Psychol. 2012;8:345-79. doi: 10.1146/annurev-clinpsy-032511-143104. Epub 2011 Dec 6. PMID 22149480
- [Background] Sanders MR, Kirby JN, Tellegen CL, Day JJ. The Triple P-Positive Parenting Program: a systematic review and meta-analysis of a multi-level system of parenting support. Clin Psychol Rev. 2014 Jun;34(4):337-57. doi: 10.1016/j.cpr.2014.04.003. Epub 2014 Apr 26. PMID 24842549
- [Background] Spijkers W, Jansen DE, Reijneveld SA. Effectiveness of Primary Care Triple P on child psychosocial problems in preventive child healthcare: a randomized controlled trial. BMC Med. 2013 Nov 11;11:240. doi: 10.1186/1741-7015-11-240. PMID 24207163
- [Background] World Health Organization (WHO). (2006). Preventing Child Maltreatment: a guide to taking action and generating the evidence. Geneva, Switzerland: World Health Organization.

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT04702191/SAP_000.pdf